CLINICAL TRIAL: NCT01244724
Title: Lexapro for Major Depression in Patients With Epilepsy
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Unable to recruit targeted #
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Forest Laboratories (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LXP-MD-109
Record Dates: First submitted 2010-11-18; First posted 2010-11-19 (Estimated); Results first posted 2015-08-03 (Estimated); Last update posted 2018-07-11 (Actual); Status verified 2018-06

CONDITIONS: Major Depression; Epilepsy
MeSH Terms: conditions — Depressive Disorder, Major; Epilepsy | interventions — Escitalopram

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lexapro (Experimental): escitalopram 10 mg or 20 mg/d
  Interventions: Drug: Lexapro

INTERVENTIONS:
Drug: Lexapro — Escitalopram will begin at 10mg. a day. Visits will occur biweekly for 12 weeks. Subjects with minimal or no response and minimal or no side effects after 4 weeks will have the dose increased to 20mg. a day. The maximum dose of escitalopram will not exceed the FDA-approved maximum dose of 20 mg per day.
  Other Names: Escitalopram

SUMMARY:
The primary objective will be to pilot the use of escitalopram for the treatment of major depression in patients with epilepsy. The secondary objectives will be to determine effect sizes on scales measuring depressive symptoms, physical symptoms, psychosocial function and quality of life, and to evaluate safety in the population of patients with epilepsy.

These results will be used to evaluate the possibility of a future double-blind, placebo controlled RCT of escitalopram for the treatment of major depression in patients with epilepsy.

DETAILED DESCRIPTION:
Rationale:

Epilepsy is a chronic disorder that adversely affects social, vocational, and psychological functioning. Despite the variety and complexity of the negative clinical associations with epilepsy, depression is remarkable in prevalence and related adverse effects on health status. An estimated 30-50% of persons with refractory epilepsy have major depression, and depression has a stronger correlation than seizure rate with quality of life. Suicide is one of the leading causes of death in epilepsy. Available data indicate that depression may result from underlying brain dysfunction rather than social and vocational disability. Most patients with depression are not screened systematically for the diagnosis, and are subsequently not treated. Although the density of serotonin receptors is greatest in limbic brain regions commonly involved in human epilepsy, such as the mesial temporal and prefrontal areas, no prior randomized controlled trials have evaluated the efficacy of serotonin reuptake inhibitors for depression in epilepsy.

Escitalopram may be an ideal SSRI for patients on antiepileptic medications because of the lack of pharmacokinetic drug interactions, which can be expected, for example, with fluoxetine or paroxetine.

Study Hypothesis:

Epilepsy patients having major depression will improve significantly over the course of a 12-week trial with escitalopram. Significant improvement will occur in ratings of depressive symptoms, physical symptoms and measures of psychosocial function and quality of life.

Primary and Secondary objectives:

The primary objective will be to pilot the use of escitalopram for the treatment of major depression in patients with epilepsy. The secondary objectives will be to determine effect sizes on scales measuring depressive symptoms, physical symptoms, psychosocial function and quality of life, and to evaluate safety in the population of patients with epilepsy.

These results will be used to evaluate the possibility of a future double-blind, placebo controlled RCT of escitalopram for the treatment of major depression in patients with epilepsy.

Study design:

An open-label design is proposed because this would be the first study of escitalopram for the treatment of major depression in patients with epilepsy.

Treatment:

Psychiatric evaluations will be done by Dr. Kocsis, who will also monitor subjects for improvement psychiatrically, as well as for potential adverse events such as agitation, psychosis, and suicidality. Subjects who are noted to have an exacerbation in their depression or develop suicidal ideation or mania may have the medication stopped or changed, based on clinician judgement. SCID assessments will be done by Dr. Bleiberg.

Escitalopram will begin at 10mg. a day. Visits will occur biweekly for 12 weeks. Subjects with minimal or no response and minimal or no side effects after 4 weeks will have the dose increased to 20mg. a day. The maximum dose of escitalopram will not exceed the FDA-approved maximum dose of 20 mg per day.

Safety Monitoring:

Safety monitoring for seizure worsening during the study will consist of the following:

Subjects will be evaluated by the study neurologist prior to starting escitalopram for a complete seizure history, and a neurologic and general physical examination. Anti-epileptic drug (AED) levels will be obtained at this baseline visit as well. The seizure count for all seizure types for the previous month will be documented. A seizure severity score for each seizure type using the National Hospital Seizure Severity Scale will be documented. Subjects will be counseled to take all AEDs regularly. After escitalopram is started, subjects will be seen every 4 weeks (3 visits) by the neurologist for a brief visit, during which an interim seizure and medical history will be obtained, and a brief neurologic examination will be performed. Seizure counts and seizure severity will be obtained for each seizure type and compared to baseline. If there is a doubling of seizure counts compared to baseline of any seizure type over any month period, the subject will be discontinued from the study and escitalopram will be discontinued. Any lesser degree of increased seizure frequency or worsened seizure severity during escitalopram treatment will prompt discontinuation of the study depending on the judgement of the investigators.

Primary and secondary efficacy measures:

Clinically rated outcomes will be the HAM-D and the CGI, which assess depressive symptoms, physical symptoms and severity of the depressive syndrome.

Self-rated assessments will include the IDS-SR for depressive symptoms, the SAS-SR for social/vocational function and the Q-LES-Q for quality of life.

Safety assessments will include hematology, chemistries, AED levels, pregnancy testing and urine drug screening prior to treatment. Hematology and chemistries, and AED levels will be repeated at week 12 or termination.

Vital signs and adverse events will be systematically recorded at each visit. Occurrence of seizures will be systematically logged during the course of the trial.

Anticipated findings:

The Wilcoxon signed-rank test will be applied to the mean scores available at weeks-1 and 0 vs. weeks 10 and 12 for the HAM-D, IDS-SR, SAS-SR and Q-LES-Q respectively. We anticipate that there will be significant differences in clinician-rated depressive symptoms and self-rated social function and quality of life from pre- to post-escitalopram treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients will be 20 males or females above the age of 18 with a current major depressive episode, as defined by DSM-IV and assessed on the MINI, of at least 4 weeks duration.
2. All subjects must have epilepsy, defined as the recurrence of seizures that are unprovoked and unpredictable, requiring treatment with an anti-epileptic medication under the care of a neurologist.
3. Subjects must be stabilized on their antiepileptic drug (AED) regimen for the previous 2 months.
4. If a vagus nerve stimulator is in place, the settings must be unchanged for the previous 2 months.
5. Patients must be ages 18 - 75 and have a 24 item Hamilton Depression Rating Scale Score (HAM-D) at intake >/= 20.
6. Subjects must be fluent in English and have the capacity to understand the nature of the study and sign the written informed consent.

Exclusion Criteria:

1. Axis II diagnosis of antisocial, schizotypal or severe borderline personality disorder(defined as patients who are high risk for being unable to complete the study due to hospitalization, suicide attempts, significant self-mutilation, or other self-injurious or destructive behavior).
2. History of psychosis, mania or hypomania.
3. Subjects with more than 10 seizures per month that involve impairment of consciousness, such as complex partial or generalized seizures.
4. Subjects unable to count seizures accurately, or do not have a someone in their home who can count seizures accurately .
5. Unstable medical or neurological disorder (other than epilepsy).
6. Epilepsies related to a progressive neurologic disease such as a brain tumor.
7. Substance abuse including ETOH within the past 6 months.
8. Need for concurrent psychotropic drugs with the exception of AEDs or zolpidem for sleep.
9. Concurrent or recent (within 3 months) entry into a new psychotherapy.
10. Actively or acutely suicidal.
11. Failure to respond to escitalopram or to two or more other adequate antidepressant trials in the past year.
12. Pregnancy or lactation.
13. Females of child bearing potential who do not practice adequate contraception.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2007-10; Primary Completion 2011-12 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Kocsis, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 26 subjects enrolled only 17 actually returned and began medication.
Period: Overall Study
Arm/Group | Lexapro
Started | 17 (Of these 15 returned for a week 2 visit and are included in the efficacy analysis.)
Week 2 Visit | 15
Completed | 9
Not Completed | 8

BASELINE CHARACTERISTICS:
Arm/Group | Lexapro
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.9 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 15
Hamilton Depression Scale [Mean (Standard Deviation); unit: units on a scale] — total score of Hamilton Depression Scale ranges from 0 (no depression) to 60 (worst depression possible)
  units on a scale | 25.5 (5.7)

OUTCOME MEASURES:

1. Primary Outcome: Hamilton Depression Scale
Description: Measure of severity of depression -total score of Hamilton Depression Scale ranges from 0 (no depression) to 60 (worst depression possible)
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Lexapro
Number analyzed (Participants) | 15
units on a scale | 13.3 (9.7)

2. Secondary Outcome: National Hospital Seizure Severity Scale
Description: Seizure severity score for each seizure type.
Time Frame: 12 Weeks
Population: Due to early termination of this study, data were not collected.
Arm/Group | Lexapro
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Twelve weeks.
Description: Adverse events were identified though standardized questionnaire administered by the research team and reviewed by the Principal Investigator.
Arm/Group | Lexapro
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 4/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lexapro (N=15)
headache (Nervous system disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No